CLINICAL TRIAL: NCT01936363
Title: Phase II Randomized Double Blind Placebo Controlled Trial of Combination of Pimasertib With SAR245409 or of Pimasertib With SAR245409 Placebo in Subjects With Previously Treated Unresectable Low Grade Ovarian Cancer
Brief Title: Trial of Pimasertib With SAR245409 or Placebo in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 200066_012; 2013-000902-40 (EudraCT Number)
Record Dates: First submitted 2013-08-23; First posted 2013-09-06 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Pimasertib; Placebo; SAR245409
MeSH Terms: conditions — Ovarian Neoplasms | interventions — XL765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pimasertib (once daily) plus SAR245409 (Experimental)
  Interventions: Drug: Pimasertib once daily; Drug: Pimasertib placebo; Drug: SAR245409
- Pimasertib (twice daily) plus SAR245409 placebo (Experimental)
  Interventions: Drug: SAR245409 placebo; Drug: Pimasertib twice daily

INTERVENTIONS:
Drug: Pimasertib once daily — Pimasertib administered as oral capsule at a dose of 60 milligram (mg) once daily until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
  Arms: Pimasertib (once daily) plus SAR245409
Drug: Pimasertib placebo — Placebo matching Pimasertib administered once daily in evening until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
  Arms: Pimasertib (once daily) plus SAR245409
Drug: SAR245409 placebo — Placebo matching SAR245409 administered once daily in morning until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
  Arms: Pimasertib (twice daily) plus SAR245409 placebo
Drug: SAR245409 — SAR245409 administered as oral capsule at a dose of 70 milligram (mg) once daily until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
  Arms: Pimasertib (once daily) plus SAR245409
Drug: Pimasertib twice daily — Pimasertib administered as oral capsule at a dose of 60 milligram (mg) twice daily until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
  Arms: Pimasertib (twice daily) plus SAR245409 placebo

SUMMARY:
This is a double blind, randomized, placebo-controlled, 2-arm, Phase 2 trial investigating the efficacy and safety of combination therapy of pimasertib plus SAR245409 and pimasertib placebo administered once per day compared to pimasertib administered twice per day plus SAR245409 placebo administered once per day in participants with previously treated unresectable low-grade serous ovarian or peritoneal carcinoma or serous borderline ovarian or peritoneal tumors.

ELIGIBILITY:
Inclusion Criteria:

* The female participant had a diagnosis of one of the following: a) low-grade serous ovarian or peritoneal carcinoma, or grade 1 serous ovarian or peritoneal carcinoma or well-differentiated serous ovarian or peritoneal carcinoma or b) serous borderline ovarian or peritoneal tumor, ovarian or peritoneal tumor of low-malignant potential, ovarian or peritoneal atypical proliferative serous tumor that recurs as low grade serous carcinoma or has invasive peritoneal implants
* The participant had at least one prior line of systemic therapy and had a tumor, which was not amenable to potentially curative surgical resection
* The participant had measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* The participant had read and understood the written informed consent form (ICF) and was willing and able to gave informed consent, fully understood the requirements of the trial and was willing to comply with all trial visits and assessments, including completion of patient-reported measures. Consent must be given before any trial related activities
* Women of childbearing potential must had a negative serum pregnancy test at the screening visit
* Women of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 2 weeks prior to screening, during and at least 3 months after the last dose of trial medication
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* The participant had previously been treated with a PI3K inhibitor and taken off treatment due to treatment related AEs
* The participant had been previously treated with a Mitogen-activated protein/extracellular signal-regulated kinase (MEK) inhibitor
* Any anti-cancer therapy or treatment incorporating chemotherapy, immunotherapy, hormonal therapy, or biologic therapy within 28 days of the start of trial treatment or within 5 times the half-life of such treatment, whichever was shorter. Treatment with nitrosoureas or mitomycin C were exceptions to this for which a treatment interval of at least 6 weeks was required
* The participant had not recovered from toxicity due to prior therapy to baseline level or National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) Grade 1 or less (except alopecia). Residual chemotherapy-induced neuropathy grade less than equal to (<=) 2 was permitted
* The participant had poor organ and marrow function as defined in the protocol
* The participant had creatine phosphokinase (CPK) elevation NCI CTCAE grade greater than equal to (>=) 2, and/or a previous history of myositis or rhabdomyolysis
* The participant had difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the trial drug. Participants requiring total parenteral nutrition were to be excluded
* The participant had a history of delayed healing/open wounds or diabetic ulcers
* The participant had a history of congestive heart failure, unstable angina, myocardial infarction, cardiac conduction abnormalities including Fridericia corrected QT interval (QTcF) prolongation of > 480 milliseconds (ms) or a pacemaker, clinically relevant impaired cardiovascular function (New York Heart Association (NYHA) class III/IV) or stroke within 3 months prior to enrollment
* The participant had a history of retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), uveitis or retinal vein occlusion (RVO), or had other relevant abnormalities identified on screening ophthalmologic examination, which might increase the risk of serous retinal detachment (SRD) or RVO
* The participant had a history of uncontrolled intercurrent illness including but not limited to an active infection, hypertension, or uncontrolled diabetes (e.g. glycosylated hemoglobin >= 8 percent [%]) that would limit compliance with treatment requirements
* Any previous malignancy treated with curative intent and the participant had been disease free for less than 5 years prior to randomization, with exception of carcinoma-in-situ of the cervix, squamous carcinoma of the skin, basal cell carcinoma of the skin
* Other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (31):
- United States (16):
  - Research site, Augusta, Georgia
  - Research site, Chicago, Illinois
  - Research site, Indianapolis, Indiana
  - Research site, Silver Spring, Maryland
  - Research site, Boston, Massachusetts
  - Research site, Ann Arbor, Michigan
  - Research site, Detroit, Michigan
  - Research site, Kansas City, Missouri
  - Research site, St Louis, Missouri
  - Research site, Kalispell, Montana
  - Research site, New York, New York
  - Research site, Cincinnati, Ohio
  - Research site, Columbus, Ohio
  - Research site, Middletown, Ohio
  - Research site, Nashville, Tennessee
  - Research site, Houston, Texas
- Australia (3):
  - Research site, Northmead, New South Wales
  - Research site, Greenslopes, Queensland
  - Research site, Subiaco, Western Australia
- Belgium (2):
  - Research site, Kortrijk
  - Research site, Leuven
- Canada (4):
  - Research site, Hamilton, Ontario
  - Research site, Toronto, Ontario
  - Research site, Montreal, Quebec
  - Research site, Québec
- Research site, Bordeaux, Gironde, France
- Research site, Chorzów, Poland
- Spain (4):
  - Research site, Palma Mallorca, Balearic Islands
  - Research site, Madrid
  - Research site, Seville
  - Research site, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participants (informed consent): Sep 2013/Oct 2014. Clinical data cut off: Jan 2018.
Groups:
- Pimasertib (Once Daily) Plus SAR245409: Participants received Pimasertib oral capsule at a dose of 60 milligram (mg) once daily along with SAR245409 oral capsule at a dose of 70 mg once daily and placebo matching to pimasertib in evening until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
- Pimasertib (Twice Daily) Plus SAR245409 Placebo: Participants received pimasertib oral capsule at a dose of 60 mg twice daily along with placebo matching to SAR245409 once daily in morning until disease progression, death, intolerable toxicity or withdrawal of informed consent, whichever came first.
Period: Overall Study
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to Treat (ITT) analysis set included all participant who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (14.07) | 50.6 (16.39) | 49.0 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Objective tumor response was defined as the presence of at least one Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to more than (<) 10 millimeter (mm). Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization until disease progression or death assessed every 8 weeks up to week 32, and thereafter every 12 weeks up to 52 months
Population: ITT analysis set included all participants who had been randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 12.5 [3.5 to 29.0] | 12.1 [3.4 to 28.2]

2. Secondary Outcome: Progression-Free Survival
Description: PFS defined as time from randomization to first documentation of objective tumor progression.CR:Disappearance of all target lesions.Any pathological lymph nodes(whether target or non-target)must have reduction in short axis to<10 mm.PR:At least 30% decrease in sum of diameters of target lesions,taking as reference baseline sum diameters.PD:At least a 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study.In addition to relative increase of 20%,the sum also demonstrate absolute increase of at least 5 mm.SD:Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,taking as reference smallest sum diameters while on study. PFS calculated as(Months)=first event date minus randomization or first dose date plus 1.Median PFS was computed using Kaplan-Meier estimates (product-limit estimates) and was presented with 95% confidence interval.The confidence intervals for median was calculated according to Brookmeyer and Crowley.
Time Frame: Time from randomization until first observation of progressive disease or death, assessed up to 52 months
Population: ITT analysis set included all participants who had been randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 32 | 33
months | 9.99 [3.42 to 15.21] | 12.71 [4.21 to NA] — The upper limit of 95% Confidence Interval for PFS could not be calculated because this upper limit was not reached due to limited number of events.

3. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control as per RECIST v.1.1 was defined as the proportion of participants with stable disease (SD), for at least 16 weeks, PR or CR according to RECIST v1.1 criteria. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: At least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Randomization until disease progression or death assessed every 8 weeks up to week 32, and thereafter every 12 weeks up to 52 months
Population: ITT analysis set included all participants who had been randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 32 | 33
percentage of participants | 50.0 [31.9 to 68.1] | 39.4 [22.9 to 57.9]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time (in months) from randomization to death. Data has been presented in terms of number participants who died and number of censored participants.
Time Frame: Time from randomization until death, assessed up to 52 months
Population: ITT analysis set included all participants who had been randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 32 | 33
Participants
  Number of deaths | 8 | 6
  Number for censored | 24 | 27

5. Secondary Outcome: Health Related Quality of Life (HrQoL) Assessed Using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item questionnaire comprising of five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact), and a global quality of life (QoL) scale summarized from two 7-point scales (overall QoL and overall general health). Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and the individual single-items ranged in score from 0 to 100. A high scale score represents a higher response level. High score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time Frame: Baseline up to disease progression or withdrawal, assessed up to 52 months
Population: Data was not collected for this outcome because as per Protocol Amendment 4 (dated 13 March 2015), the collection of patient-reported health-related quality of life outcomes was discontinued.
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Health Related Quality of Life (HrQoL) Assessed Using European Organization for Research and Treatment of Cancer (EORTC) Ovarian-Specific Module Quality of Life Questionnaire Ovarian Cancer Module (QLQ-OV28)
Description: EORTC QLQ-OV28 assesses disease and treatment-related symptoms of ovarian cancer. The 28-item module comprises of 6 symptom scales (abdominal/gastrointestinal symptoms, peripheral neuropathy, other chemotherapy side-effects, hormonal symptoms, body image, attitude to disease and treatment), and sexual functioning. All of the scales and the individual single-items ranged in score from 0 to 100. Higher scores indicate a better quality of life.
Time Frame: Baseline up to disease progression or withdrawal, assessed up to 52 months
Population: as for outcome 5
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation of Treatment and Death
Description: TEAEs, Serious TEAEs and AEs were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0. An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A Serious Adverse Event was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to data cut-off that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: First dose of study drug up to 52 months
Population: Safety population (SAF) analysis set included all participants who received at least one dose of any trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 32 | 32
Participants
  TEAE | 32 | 32
  Serious TEAE | 16 | 18
  TEAE leading to discontinuation of study treatment | 16 | 12
  Death | 2 | 3

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Dose of Pimasertib and SAR245409
Time Frame: Pre-dose Hour 0.5, 1.5, 4.5 8 post dose on Day 15, 29, 43
Population: As per changed in planned analysis the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Area Under the Curve (AUC) After Dose of Pimasertib and SAR245409
Time Frame: Pre-dose Hour 0.5, 1.5, 4.5 8 post dose on Day 15, 29, 43
Population: As per changed in planned analysis the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Molecular Alterations in MAPK and/or PI3K Signaling Pathway Components/Modulators in Tumor Tissue and Blood
Time Frame: Screening visit (day -28 to 1)
Population: As per changed in planned analysis the outcome measure related to pharmacodynamics parameters was not assessed.
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 52 months
Description: SAF included all participants who received at least 1 dose of any trial treatment. SAF for "Pimasertib (Once Daily) Plus SAR245409" = 32 participants and "Pimasertib (Twice Daily) Plus SAR245409 Placebo" = 32 participants. Adverse events analysis was based on the SAF which includes 64 participants but 1 participant was randomized by error and not treated therefore not adverse event analysis.
Arm/Group | Pimasertib (Once Daily) Plus SAR245409 | Pimasertib (Twice Daily) Plus SAR245409 Placebo
Serious Adverse Events (participants affected / at risk) | 16/32 | 18/32
Other Adverse Events (participants affected / at risk) | 32/32 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib (Once Daily) Plus SAR245409 (N=32) | Pimasertib (Twice Daily) Plus SAR245409 Placebo (N=32)
Cardiac arrest (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Intraocular pressure increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 2 | 0
Device related infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib (Once Daily) Plus SAR245409 (N=32) | Pimasertib (Twice Daily) Plus SAR245409 Placebo (N=32)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Vision blurred (Eye disorders) | 16 | 11
Macular detachment (Eye disorders) | 6 | 5
Visual impairment (Eye disorders) | 7 | 3
Retinal detachment (Eye disorders) | 3 | 6
Eyelid oedema (Eye disorders) | 2 | 4
Subretinal fluid (Eye disorders) | 1 | 2
Visual acuity reduced (Eye disorders) | 1 | 2
Eye disorder (Eye disorders) | 2 | 0
Periorbital oedema (Eye disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 26
Nausea (Gastrointestinal disorders) | 22 | 13
Vomiting (Gastrointestinal disorders) | 16 | 14
Stomatitis (Gastrointestinal disorders) | 13 | 9
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Constipation (Gastrointestinal disorders) | 6 | 5
Dry mouth (Gastrointestinal disorders) | 8 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Abdominal distension (Gastrointestinal disorders) | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 19 | 14
Oedema peripheral (General disorders) | 11 | 15
Pyrexia (General disorders) | 6 | 8
Chills (General disorders) | 9 | 2
Asthenia (General disorders) | 0 | 8
Face oedema (General disorders) | 4 | 3
Peripheral swelling (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 5 | 8
Conjunctivitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 19 | 19
Aspartate aminotransferase increased (Investigations) | 7 | 4
Alanine aminotransferase increased (Investigations) | 7 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Weight increased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 11 | 7
Headache (Nervous system disorders) | 3 | 6
Paraesthesia (Nervous system disorders) | 5 | 2
Dysgeusia (Nervous system disorders) | 2 | 3
Migraine (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 5 | 0
Dysuria (Renal and urinary disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 2
Dry eye (Eye disorders) | 2 | 0
Mass (General disorders) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 1
Tremor (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 1 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other